CLINICAL TRIAL: NCT02240329
Title: Assessment of Dystussia in Traumatic Brain Injury
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 217-2012
Record Dates: First submitted 2014-06-05; First posted 2014-09-15 (Estimated); Results first posted 2015-10-28 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-09

CONDITIONS: TBI; Brain Injury
Keywords: respiratory; cough
MeSH Terms: conditions — Brain Injuries; Cough | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Individuals with TBI (Other): Individuals who have sustained a traumatic brain injury during the previous five years. Will have the following tests performed: Neuropsychological Testing and Measures of TBI severity; Cough and respiratory measures (including Maximum Respiratory Pressures); and Capsaicin cough sensitivity testing.
  Interventions: Behavioral: Neuropsychological Testing and Measures of TBI severity; Behavioral: Respiratory measures; Drug: Capsaicin cough sensitivity testing

INTERVENTIONS:
Behavioral: Neuropsychological Testing and Measures of TBI severity — A brief cognitive assessment will be given to each participant when he or she presents for this project.
Behavioral: Respiratory measures — We will collect measures of cough airflow and breathing strength.
Drug: Capsaicin cough sensitivity testing — Subjects will inhale a saline vapor mixed with various concentrations of capsaicin powder in order to determine how sensitive his or her cough response is.
  Other Names: Cough reflex testing

SUMMARY:
The purpose of this research study is to evaluate coughing in people who have had a brain injury. It is hypothesized that individuals who have sustained a brain injury will demonstrate differences in cough waveform and respiratory measures compared to individuals who have not sustained a brain injury.

DETAILED DESCRIPTION:
Recovery of people with mild, moderate, or severe swallowing, speech, hearing, and cognitive-communication impairments is best facilitated by a team of multidisciplinary specialists. Symptoms associated with traumatic brain injury (TBI) include disordered swallowing (dysphagia), ataxia and, frequently, but not inevitably, dysarthria or disorder of speech. Airway compromise also exists in the form of impaired cough, or dystussia. In view of the frequency of oral intake problems in individuals with TBI and the presence of weakened cough, or absence of cough, along with the added challenge of the cognitive-communicative problems, further studies are needed to increase our understanding of the degree of disordered airway protection. From this work appropriate intervention strategies can be designed along with an understanding of the compensations that may be used to assist with improving swallow and airway safety, oral intake and management.

Informed Consent Process:

Investigators working with subjects with TBI, and who are also aware of this study, will have the ability to provide potential participants with a business card containing only the name of the study coordinator (Dr. Erin Silverman) as well as her email and telephone numbers. The individual participants will be responsible for contacting Dr. Silverman if they wish to participate. Additional participants will be recruited via face to face methods and by the previously IRB-approved study flyer at local brain injury support groups and Shands Rehabilitation Hospital.The staff member consenting (Dr. Silverman) has completed University of Florida training on HIPAA and privacy issues. Subjects do not have to give an immediate response about enrolling and may freely discuss the study with people of their choice before making a decision. Capacity to consent will be decided by the consenting staff member (Dr. Silverman). The study will be explained to the subject, any questions answered, and a written and signed consent completed along with a HIPAA authorization. Written consent will be obtained prior to collection of any health history or study data. Once written informed consent is obtained, Dr. Silverman will conduct an extensive interview in order to insure the subject meets all required inclusionary/exclusionary criteria.

Neuropsychological Testing: The MOCA (Montreal Cognitive Assessment) will be administered by Dr. Silverman, on each participant, upon entry into the study.

Measures of TBI severity: Multiple studies have correlated severity of TBI upon initial admission related to the TBI with swallowing function. The Glasgow Coma Scale (GCS) and Rancho Los Amigos Scale (RLAS) are commonly administered upon admission of TBI patients. When available (availability may vary depending on the hospital at initial admission) we will record the GCS and/or RLAS scores from admission. As well, the investigators will administer the RLAS upon enrollment in the study. These measures will be incorporated into our statistical model to better understand the heterogeneity of cognitive impairment on swallow and cough function.

Cough and respiratory measures: Pulmonary status screening measures: The forced expired volume in the first second (FEV1) of a forced vital capacity (FVC) exhalation are measures used to screen pulmonary function (American Thoracic Society). Spirometry is used to derive FVC, FEV1 and the ratio FEV1/FVC measures (Spirovision 3+m, Futuremed). Alternatively, if the subject is unable to perform the cognitive voluntary spirometric task, upper airway respiratory resistance will be measured with impulse oscillometry (lOS, Jaeger Instruments).

Maximum Respiratory Pressures: Maximum inspiratory and expiratory pressures are an indirect measure of inspiratory and expiratory muscle strength, respectively. The ability to generate high expiratory airflows is essential to producing high expiratory airflow, and subsequently cough production and will be measured at the initial assessment in all studies.

Cough: The participant will be instrumented for the measurement of the respiratory airflow pattern during spontaneous breathing, voluntary cough and reflex capsaicin induced cough. A facemask with a pneumotachograph will be used to record the airflow changes associated with spontaneous breathing and cough. The mouth airflow signal will be digitized and recorded on a desktop computer (Chart, ADinstruments, Inc). Inspiratory and expiratory muscle EMG will be recorded to provide a neuromuscular motor assessment of cough strength. The computer signals will be analyzed to determine inspiratory breath phase, expiratory breath phase, inspiratory cough phase, cough compression phase, and expiratory cough phase. Because it has been reported that brain injury differentially affects the neuromuscular motor pattern of voluntary and reflex elicited coughs, it is essential to elicit coughs with both peripheral afferent stimulation (capsaicin; reflexive cough) and voluntary induced cough in these TBI participants.

Capsaicin administration: After the participant is instrumented with the facemask, he/she will be seated comfortably in a chair in front of an airflow fume hood. The airflow fume hood prevents exposure of the participant and experimenter to the nebulized solution except when the participant inhales for the capsaicin challenge. Participants will inspire deeply through the nebulizer (containing the capsaicin or a vehicle solution) coupled to the facemask and pneumotachograph. The outflow nebulizer gas will be passed through an isopropyl alcohol solution to remove capsaicin from the air vented into the fume hood. Cough threshold and sensitivity will be determined using our established randomized block presentation method of graded capsaicin concentrations (0-2001-JM). The investigators have an FDA IND # 76866 for the use of capsaicin in the study of cough motor pattern. This will take 10-15 minutes to complete.

Design and Procedures: This project will address the Specific Aim over a 1-year time period. Our Specific Aim will focus on characterizing the mechanical features of swallow and cough motor function in subjects with TBI and the swallow and cough reconfiguration of respiratory pattern. Our Specific Aim will allow us to determine the relationship between TBI and both swallow and cough dysfunction.

Study Protocol: Subjects with a medical history of TBI will be recruited from community TBI support groups and through face to face recruitment procedures. Once informed consent has been obtained, relevant medical history will be reviewed, and the participants will complete screening procedures to determine inclusionary/exclusionary criteria. If inclusionary and exclusionary criteria are met, participants will complete the following tests:

* MIP and MEP measurement
* Reflex and voluntary cough assessments

Timeframe: This is a one-time visit study. Therefore, participants will be followed only on the day they present for study procedures. There will be no follow up beyond this day.

ELIGIBILITY:
Inclusion Criteria:

1. TBI within 5 years - may have accompanying neck injury but not extensive reconstruction of oral structures.
2. Pulmonary function screening: FEV1 >75%, FVC > 75% and FEV1/FVC ratio of >75% of age, sex and ethnicity corrected predicted values, impulse oscillometry R5 resistance measurement within 15% of age, sex and ethnicity corrected predicted values.
3. Medical status permits participation.
4. Cognitive status permits participation.

Exclusion Criteria:

1. Refuses consent.
2. Cognitively incapable of informed consent
3. Active substance dependence/use (from clinical interview/record review)
4. Diagnosis of moderate to very severe chronic obstructive pulmonary disease (COPD; from patient interview)
5. History of chronic cough and/or cough syncope (From clinical interview)
6. History of cancer in the head or neck (From clinical interview)
7. History of radiation to the head or neck (From clinical interview)
8. History of stroke or other neurodegenerative disease (From clinical interview) Participants will be enrolled without regard for sex, ethnicity, or age.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2013-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul W Davenport, Ph.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Silverman E, Sapienza CM, Miller S, Carnaby G, Levy C, Tsai HW, Davenport PW. Preliminary Evidence of Reduced Urge to Cough and Cough Response in Four Individuals following Remote Traumatic Brain Injury with Tracheostomy. Can Respir J. 2016;2016:6875210. doi: 10.1155/2016/6875210. Epub 2016 Sep 27. PMID 27774033

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Individuals With TBI
Started | 4
Determination of Urge to Cough | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Individuals With TBI
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.38 (13.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Average Urge to Cough (UTC) Following Administration of 200 Micro Mole Capsaicin Solution Concentration
Description: Following 30 seconds of tidal breathing (to allow for acclimation to the facemask), participants were instructed to "take a sharp breath in" whereupon the nebulized capsaicin solution was automatically administered by the dosimeter. Following each aerosol presentation, the participant was instructed to rate their UTC using a modified Borg Rating Scale where 1 = no UTC and 10 = maximum UTC. Between presentations, participants were given a minimum of a one-minute rest period where they were offered water. An average across all measurements was performed for the analysis.
Time Frame: Day 1
Measure: Mean (Standard Error); unit: Units on a Borg scale
Arm/Group | Individuals With TBI
Number analyzed (Participants) | 4
Units on a Borg scale | 4.5 (1.68)

2. Primary Outcome: Number of Coughs in Response to Stimulation With 200 Micro Moles Capsaicin in Solution
Description: The total cough count (CTot) was determined by counting all cough events that occurred following each presentation of capsaicin solution. CTot was made, in real time, by two investigators and confirmed via review of the recorded cough airflow signal. Capsaicin concentration necessary to elicit a two cough threshold response (C2) within 30 seconds of presentation, on at least two (out of three) trials of that concentration, was identified from the cough count record. An average across all measurements was performed for the analysis.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: cough events following stimulation
Arm/Group | Individuals With TBI
Number analyzed (Participants) | 4
cough events following stimulation | 2.83 (0.43)

ADVERSE EVENTS:
Time Frame: Duration of study (one day)
Arm/Group | Individuals With TBI
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No